CLINICAL TRIAL: NCT06652919
Title: Development and Validation of Materials for the Pharmaceutical Care of Organ Transplant Recipients in Community Pharmacy: Survey on the Evaluation of Medication Information Leaflets for Organ Transplant Patients
Brief Title: Survey on the Evaluation of Medication Information Leaflets for Organ Transplant Patients
Status: Recruiting | Type: Observational
Sponsor: Universität Münster (Other)
Responsible Party: Principal Investigator, Li-Yun Chen, Principal Investigator, Universität Münster
Other Study IDs: Clinical Pharmacy Uni MS_2024
Record Dates: First submitted 2024-10-16; First posted 2024-10-22 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Organ Transplantation
Keywords: Organ transplantation; Consumer Information Rating Form; Pharmaceutical Care; Community Pharmacy; Patient Information Leaflets

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to collect feedback from organ transplant patients or their caregivers/relatives on the medication information leaflets we've developed, using a questionnaire, and to adjust the content to better meet the specific needs of this unique patient group.

DETAILED DESCRIPTION:
Introduction:

Organ transplantation is a life-saving procedure, but it also marks the beginning of a lifelong journey for patients. In 2023 alone, over 3,600 organ transplants were performed in Germany, with kidney, liver, heart, and lung transplants being the most common. Following a transplant, patients must take a combination of immunosuppressive medications to prevent their body from rejecting the new organ. These drugs, while essential, come with significant risks. Many of which have a very narrow therapeutic range and a high risk of drug interactions. Additionally, these medications have unique side effects that can affect mortality and health-related quality of life (HRQOL). As a result, organ transplant patients require constant medical monitoring and comprehensive education about their medications to ensure long-term graft survival and a better quality of life.

Community pharmacies in Germany have recognized the need to support these patients. Since 2022, community pharmacies have been offering pharmaceutical care services specifically tailored to organ transplant recipients, focusing on safe medication use and personalized counseling, including brown-bag reviews. This service is covered by health insurance and aims to reduce administration errors, improve therapy adherence, and enhance overall patient safety. However, despite nearly 4,000 new organ transplants each year, only a small fraction of these patients-less than 3%-benefit from these services annually. The reality is that public pharmacies rarely interact with transplant patients, as they make up a small group. Furthermore, there is currently a lack of adequate materials to support the provision of this service for transplant patients.

This research project addresses this gap by developing and validating specific materials that will help pharmacies deliver high-quality pharmaceutical care to organ transplant recipients. A key element of this project is the medication information leaflets designed by the investigators, which aim to enhance patients' understanding of their immunosuppressive therapy, reduce medication use errors, and ultimately improve medication safety.

The aim of this study is to collect feedback from organ transplant patients or their caregivers/relatives on these medication leaflets, using a questionnaire instrument called "Adapted Consumer Information Rating Form (CIRF)", developed by Krass et al. The results will help the investigators evaluate the quality of the medication information leaflets in terms of their content and design. This will also assist the investigators in adjusting the content to better meet the specific needs of this unique patient group in the future.

Study design:

This pilot study is designed as a descriptive survey. It involves a one-time survey, either online or in paper form, that collects data on participants' evaluations and opinions regarding the medication information sheets. The instrument that is used, the original Adapted CIRF, was initially translated by the investigators through a peer review process, including cultural adaptation from English to German. After two rounds of peer review, the final version was produced. Permission for the use and translation of the original Adapted CIRF was obtained from Krass et al. Additionally, demographic data will be collected in the study. This study was approved by the Ethics Committee: Ethik-Kommission der Ärztekammer Westfalen-Lippe und der Westfälischen Wilhelms-Universität Münster.

The recruitment of the participants will be conducted through cooperating pharmacies and patient self-help groups, and participation in the questionnaire is voluntary. Data protection measures will be taken into account to ensure the confidentiality and security of participants' information.

Procedure for participation in the study:

1. The study begins as soon as the participants have agreed to the consent form.
2. The study consists of two parts. In Part 1, participants are asked to select a medication information sheet and thoroughly read it.
3. In Part 2, participants will ask to complete the questionnaire.
4. After completing the questionnaire, the participation is considered finished. The process will take approximately 10 to 20 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone solid organ transplantation (kidney, liver, heart, lung)
* Caregivers or family members of organ transplant patients
* German-speaking individuals
* adult

Exclusion Criteria:

* Individuals who are not able to provide consent
* Non-German-speaking individuals
* under 18 years old
* Patients who have undergone organ transplantation and are no longer taking immunosuppressants

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone solid organ transplantation (kidney, liver, heart, lung) or their caregivers/family members
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-11-06 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Consumer Information Rating Form (CIRF): Mean "comprehensibility" score, mean "future use" score, mean "utility" score and mean "design quality" score. | 3 months
  In this research, the measurement instrument called the Consumer Information Rating Form (CIRF) is used, though the content has been slightly adapted to fit our study. It was developed as a direct method for quantifying consumers' perceptions of written patient information, including their views on its comprehensibility, utility, and overall design quality.
  In the questionnaire, four perspectives will be evaluated using Likert scales, including "comprehensibility" (5 items, with a total score range from 5 to 25), "future use" (3 items, with a total score range from 3 to 15), "utility" (5 topics with two perspectives: the amount of information provided and its usefulness, with a total score range from 3 to 20.), and "design quality" (6 items, with a total score range from 6 to 30). Higher scores indicate better quality of the patient information leaflet.
Participants' characteristics | 3 months
  Gender, age group, highest level of education, current employment status, if participant has worked in the healthcare system, Which patient information leaflet did the participant evaluate? What type of organ transplant has the participant or the person they look after received? (Kidney, liver, heart, or lung transplant), How long has it been since the transplant?

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Pharmaceutical and Medicinal Chemistry, Clinical Pharmacy, University of Münster, Münster, North Rhine-Westphalia, Germany